CLINICAL TRIAL: NCT02623907
Title: Registry Study of Aortic Valve Diseases in Chinese Elderly
Brief Title: China Valve Registry Study-1
Acronym: CHIVAS-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHIVAS2015
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Heart Valve Diseases
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AS group: Severe AS patients, without severe AR
- AR: Severe AR patients, without severe AS

SUMMARY:
With the aging of Chinese population, degenerative valvular disease is becoming more and more frequent, which has brought a heavy burden to our society. Taking aortic stenosis (AS) as an example, the incidence of AS in population over the age of 65 are about 2%, and in population above the age of 85 can be amounted to 4-8%, in the Western country. Since the invention of transcatheter aortic valve replacement (TAVR),aortic valve disease (AVD),including AS and aortic regurgitation (AR), has attracted more and more attention. To date, there are few data about the prevalence of AVD in China. The characteristics and prognosis of AVD in China are still unknown. Therefore, the investigators design a prospective, observational cohort study to investigate characteristics, treatments and prognosis of AVD in Chinese elderly population. The results of the study will provide a basis for the future national health policy for prevention and treatment of AVD in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Severe AS or AR indicated by echocardiography ;
* 60 years old or older.

Exclusion Criteria:

* Having both Severe AR and Severe AS;
* Having underwent surgical or transcatheter treatment for AVD;
* Non-degenerative AVD.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aging more than 60 years diagnosed with severe AS or AR by echocardiography will be collected from multiple institutions.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular (CV) death or hospitalization for heart failure (HF) | 36 months
  from date of enrollment until the date of first documented HF or date of death from any cause, whichever came first, up to 36 months
Surgical or transcatheter aortic valve replacement | 36 months
  from date of enrollment until the date of surgical or transcatheter aortic valve replacement, whichever came first, up to 36 months

SECONDARY OUTCOMES:
Number of all-cause mortality | from date of enrollment until the date of death for any-cause, up to 36 months
Number of patients developing major cardiovascular and cerebral events (MACCE) | 36 moths

IPD SHARING:
Plan to Share IPD: Undecided